CLINICAL TRIAL: NCT00144235
Title: A 28 Day, Randomised, Double-blind, Placebo-controlled, Single-centre Trial to Evaluate the Efficacy and Safety of Pharmaton® PHL 00749 Film Coated Tablets (G115 40 mg, Multivitamin, Multimineral + Guarana 75 mg) 1/Day p.o. in Improving Mental Performance and to Decrease Fatigue in Healthy Male and Female Subjects in Regular Employment.
Brief Title: Pharmaton Upgrade in Improving Mental Performance and Decreasing Fatigue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1232.1
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Mental Competency; Mental Fatigue
MeSH Terms: conditions — Mental Fatigue

INTERVENTIONS:
Drug: Pharmaton PHL 00749
Drug: Placebo

SUMMARY:
To assess the efficacy and safety of Pharmaton? PHL 00749 in improving cognitive function and allevi ating mental and physical stress in healthy male and female subjects leading demanding lifestyles.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomised, parallel group trial in healthy male and fem ale subjects in regular employment. The duration of dosing will be 28 '(+/- 1)' days and assessments w ill be made on two visits (visits 2 and 3) with a training on the CDR system at the screening visit.

The subjects will receive one bottle with 35 tablets [of either Ginseng G115 40 mg, multivitamin, mu ltimineral '+' Paullinia cupana extract PC102 75 mg (Guarana) or placebo] from the pharmacy at the in vestigational site. The subjects should take the study drug from day 0 to day 28 '(+/- 1)' Subjects will be assigned to one of the two treatment groups randomly. The allocation ratio is 2:1..

Study Hypothesis:

H0: No difference exists between the treatment and the placebo groups in terms o f baseline-adjusted change in Power of Attention after 28 days and averaged over 4 and 6 hour time point. H1: A difference exists between the treatment and the placebo groups in terms of baseline-adjusted change in Power of Attention after 28 days and averaged over 4 and 6 hour time point. The null and alternative hypotheses for the secondary endpoints are set up accor dingly. The statistical testing will be carried out at the 0.05 level of signifi cance. The test will be performed two-tailed.

Comparison(s):

The comparator is a matching placebo film-coated tablet without active ingredien ts.

ELIGIBILITY:
INCLUSION CRITERIA Healthy male and female subjects in regular employment, aged between 20 and 50 y ears. Subjects who give written informed consent in accordance with GCP and local legi slation.

EXCLUSION CRITERIA Subjects who present with clinical depression. Subjects showing evidence of dementia. Clinically relevant abnormalities in medical history or examination. Subjects who have participated in a clinical study within 3 months prior to the start of the study. History of drug and/or alcohol abuse. Subjects who smoke more than 10 cigarettes per day. Subjects who in the opinion of the Investigator are heavy users of other tobacco or nicotine products (e.g. snuff, chewing tobacco, nicotine patches, nicotine g um, etc.). Subjects who have a history of food and/or drug allergies relevant to the study compound. Clinically relevant deviation from normal of any finding during pre-study medica l screening. Subjects who are unable to perform the cognitive tests. Subjects currently taking a cognition enhancing substance, including any Ginkgo, ginseng or guarana product. Any subject regularly taking a medication who might stop doing so at some time d uring the active dosing phase. Pregnant or lactating women or female subjects of child-bearing potential not us ing adequate means of birth control (condoms, contraceptive pills, IUDs, sterili sation). Subjects already taking other multi-vitamin products during the last 2 weeks. Healthy subjects who are regularly taking drugs which act on the Central Nervous System (CNS).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 412
Dates: Start 2005-03; Primary Completion 2005-07 (Actual); Study Completion 2005-07

PRIMARY OUTCOMES:
Primary Endpoint: The baseline (day 0 pre-dose) adjusted change in the CDR Factor, Power of Attention, at day 28 averaged over the 4 and 6 hour post-dosing time points. | 28 days

SECONDARY OUTCOMES:
The baseline (day 0 pre dose) adjusted change in the CDR Factor, Power of Attention, at day 0 averaged over the 4 and 6 hour post dosing time points. | 28 days
The baseline (day 0 pre-dose) adjusted change scores at day 28 in the CDR factors: Continuity of Attention, Quality of Episodic Secondary Memory, Speed of Memory and Quality of Working Memory | 28 days
The baseline (day 0 pre-dose) adjusted change scores at day 28 in the individual CDR tests. | 28 days
The baseline (day 0 pre-dose) adjusted change scores at day 0 in the CDR factors: Continuity of Attention, Quality of Episodic Secondary Memory, Speed of Memory and Quality of Working Memory. | 28 days
The baseline (day 0 pre-dose) adjusted change scores at day 0 in the individual CDR tests | 28 days
The day 0 pre-dose adjusted change scores at day 28 in the CDR factors: DailyStressInventory,Pro- and RetrospectiveMemoryQuest,CognitiveFailures quest, St. Mary's HospitalSleep Quest,SpielbergerStateTraitAnxiety Quest,PsychologicalGeneralWell-Being Quest | 28 days
Incidence of all adverse events | 28 days
Vital signs (BP and HR) | 28 days
Overall tolerability assessment by the subject and investigator | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Pharmaton
Locations (1):
- Boehringer Ingelheim Investigational Site, Aldershot, United Kingdom